CLINICAL TRIAL: NCT00893633
Title: Prospective Case-Only Study of Neuromuscular Pathology in Patients on Mechanical Ventilation in the Neurosurgical Intensive Care Unit
Brief Title: Critical Illness Neuromuscular Abnormalities in Neurocritical Care Patients
Status: Completed | Type: Observational
Sponsor: Clinical Institute of the Brain, Russia (Other)
Collaborators: City Hospital No 40, Saint Petersburg, Russia (Other)
Responsible Party: Andrey Alasheev, Clinical Institute of the Brain, Russia
Other Study IDs: CINMAs-2004
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Muscle Weakness; Critical Illness
Keywords: neuromuscular diseases; critical illness; mechanical ventilation; phrenic nerve; nerve conduction studies
MeSH Terms: conditions — Muscle Weakness; Critical Illness; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this research is to investigate critical illness neuromuscular abnormalities in neurocritical care patients.

DETAILED DESCRIPTION:
Since 1984, the problem of critical illness neuromuscular abnormalities (CINMAs) has attracted considerable interest. According to these studies, CINMAs include the muscular weakness that accompanies critical illness resulting from polyneuropathy and/or myopathy and can be seen in 25-85% of cases of critically ill patients. Clinically, CINMAs present as symmetric flaccid tetraparesis and difficulty weaning off mechanical lung ventilation. However, these data are derived from treating non-specialized intensive care unit (ICU) patients. In this research, we wished to investigate CINMAs in neurocritical care patients. From day one of the patients' participation in the research and until a discharge from the ICU (or death), daily neurological surveys and weekly nerve conduction studies were performed. Based on the results of each nerve conduction study, an index of neuromuscular damage was noted to evaluate the severity of the CINMAs. Needle electromyography and muscle biopsy were not used

ELIGIBILITY:
Inclusion Criteria:

* Age: 16 years and older
* Acute primary cerebral pathology
* Mechanical ventilation
* Signs of systemic inflammatory response
* Exclusion of the possibility of an initial pathology of the spinal cord, peripheral nervous system and muscles in past medical history

Exclusion Criteria:

* Brain stem or bilateral hemispheric lesions with tetraparesis at the onset of illness
* Inability to perform high-grade nerve conduction studies

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from neurosurgical ICU in city clinical hospital
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2004-03; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
incidence of critical illness neuromuscular abnormalities (CINMAs) | within the first week of mechanical ventilation

SECONDARY OUTCOMES:
clinical and neurophysiological characteristics of CINMAs | within the first week of mechanical ventilation
influence оf phrenic nerve pathology on weaning from mechanical ventilation | during weaning period
dynamics of the neurophysiological characteristics of CINMAs | during stay in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Andrey M Alasheev, MD, PhD, Principal Investigator — Clinical Institute of the Brain, Russia
Locations (1):
- Clinical Institute of the Brain, Yekaterinburg, Russia